CLINICAL TRIAL: NCT04799678
Title: Collecting Anonymous Voice Samples From Users of the Smart Asthma App
Brief Title: Pilot Voice Sample Collection From People With Asthma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Thomas Antalffy (Industry)
Responsible Party: Sponsor-Investigator, Thomas Antalffy, Managing Director, Smart Respiratory Products Ltd.
Organization: Smart Respiratory Products Ltd. (Industry)
Other Study IDs: VoiceRecPilot
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Asthma Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Current user of the Smart Asthma app
  Interventions: Other: Recording voice samples

INTERVENTIONS:
Other: Recording voice samples — A maximum of 9 voice sample recording session will be carried out on their phones and take less than 2 minutes each

SUMMARY:
Human speech is as unique as a fingerprint and analysing speech had advanced so much that speech can now be used instead of PIN numbers in banking.

The investigators want to find out whether changes in everyday speech can signal the worsening of asthma.

The investigators are planning to collect voice samples from people as their asthma gets better and worse in order to analyse the changes in voice quality - if any.

The participants donating the voice samples will remain anonymous and the voice files will be transferred securely to our analytic system.

DETAILED DESCRIPTION:
Over 18 users of the Smart Asthma app (by Smart Respiratory Products Ltd) will be asked if they wish to participate in the study by recording voice samples. The question will be posed within the app and can be answered with a tap.

Those interested in participating will be shown a short plain English description of the goals and methodology of the project before enrolled.

A maximum of 9 voice sample recording session will be carried out on the phones of participants and take less than 2 minutes each, so participants will spend a total of fewer than 18 minutes during the entire trial.

Sessions will be offered after participants have recorded their asthma symptoms, lung function and inhaler use in the normal course of using the app. Participants may accept or decline each individual offer to record their voice.

Participants will have a chance to play each voice recording before sharing it anonymously with the investigators. Participants can discontinue their participation at any time and can ask investigators to delete all their data.

The investigators will be analyse collected voice samples for changes in voice quality. The changes in voice quality will be compared against changes in lung function and asthma symptoms to determine what changes in voice quality, if any, are indicative of a change in asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Current user of the Smart Asthma app
* Over 18
* Volunteers to participate
* Agrees to terms

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current user of the Smart Asthma app
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in voice quality | A maximum of 9 voice sample recording session, 2 minutes each, will be carried out during the 6 months of the study
  Voice is an effective biomarker to monitor and predict the loss of asthma control

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Antalffy, MD, Principal Investigator — Managing Director

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD